CLINICAL TRIAL: NCT01224808
Title: An Open-Label, Multi-Centre Extension Study to Assess the Efficacy and Safety of Biostate® in Paediatric, Adolescent, and Adult Subjects With Von Willebrand Disease Who Completed Clinical Studies CSLCT-BIO-08-52 or CSLCTBIO-08-54
Brief Title: Extension Study of Biostate in Subjects With Von Willebrand Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-09-64; 2009-017301-11 (EudraCT Number); 1498 (Other: CSL Behring)
Record Dates: First submitted 2010-06-08; First posted 2010-10-20 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Von Willebrand Disease
Keywords: von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Biological: Biostate

INTERVENTIONS:
Biological: Biostate — Single bolus doses, administered intravenously. Frequency and dose will be determined by the Investigator based on the subjects clinical condition, previous VWF concentrate requirements, response to therapy, weight and reason for usage.

SUMMARY:
The aim of the Von Willebrand Disease (VWD) therapy is to treat and prevent bleeding episodes due to abnormal platelet adhesion and abnormal blood coagulation as a result of low or abnormal Von Willebrand Factor (VWF) and/or Factor VIII (FVIII) levels. The long-term efficacy and safety of a VWF/FVIII concentrate, Biostate, will be investigated in children, adolescents, and adults with VWD in whom treatment with a VWF product is required for prophylactic therapy, haemostatic control during surgery, or control of a non-surgical, spontaneous, or traumatic bleeding event.

ELIGIBILITY:
Inclusion Criteria:

* Have completed Study CSLCT-BIO-08-52 (Assessment of Efficacy and Safety of Biostate in Paediatric Subjects with Von Willebrand Disease) or Study CSLCT-BIO-08-54 (Assessment of Efficacy and Safety of Biostate in Adolescent or Adult Subjects with Von Willebrand Disease).
* The subject and/or his/her legal guardian understand(s) the nature of the study and has/have given written informed consent to participate in the study and is/are willing to comply with the protocol.

Exclusion Criteria:

* Early discontinuation of a subject from the main studies CSLCT-BIO-08-52 or CSLCT-BIO-08-54.
* Mental condition rendering the subject (or the subject's legal guardian) unable to understand the nature, scope and possible consequences of the study.
* Any condition that is likely to interfere with evaluation of the IMP or satisfactory conduct of the study.
* Are not willing and/or not able to comply with the study requirements.
* Employee at the study site, or spouse/partner or relative of the Investigator or Subinvestigators.
* Female subjects of childbearing potential either not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study, or not sexually abstinent for the entire duration of the study, or not surgically sterile.
* Intention to become pregnant during the course of the study.
* Pregnancy, or nursing mother.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Haemostatic efficacy | Up to 32 months

SECONDARY OUTCOMES:
Development of FVIII inhibitors | Up to 32 months
Development of VWF inhibitors | Up to 32 months
Frequency of Adverse events (AEs) per subject | 32 months
Severity of AEs per subject | 32 months
Severity of AEs per infusion | 32 months
Causality of AEs per subject | 32 months
Causality of AEs per infusion | 32 months
Frequency of Adverse events (AEs) per infusion | 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (6):
- Study Site, Sofia, Bulgaria
- Study Site, Bremen, Germany
- Poland (2):
  - Study Site, Warsaw
  - Study Site, Wroclaw
- Study Site, Barnaul, Russia
- Study Site, Lviv, Ukraine